CLINICAL TRIAL: NCT03136393
Title: A Protocol for a Cluster Randomized Controlled Trial Measuring the Effect of Dietary Counseling During Pregnancy on Infant Birthweight in Nankumba, Mangochi District, Malawi
Brief Title: Effect of Dietary Counseling During Pregnancy on Infant Birthweight in Mangochi , Malawi
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Oslo (Other)
Collaborators: University of Malawi (Other); University of Adelaide (Other); London School of Hygiene and Tropical Medicine (Other)
Responsible Party: Principal Investigator, Penjani Rhoda Kamudoni, Dr, University of Oslo
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: NFR-220895
Record Dates: First submitted 2016-03-05; First posted 2017-05-02 (Actual); Last update posted 2023-06-18 (Actual); Status verified 2023-06

CONDITIONS: Maternal Exposure During Pregnancy
Keywords: nutrition; pregnancy; birth weight
MeSH Terms: conditions — Birth Weight

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control (Active Comparator): Community based antenatal counselling
  Interventions: Behavioral: Community based antenatal counselling
- Intervention (Experimental): Community based dietary counselling
  Interventions: Behavioral: Community based dietary counselling; Behavioral: Community based antenatal counselling

INTERVENTIONS:
Behavioral: Community based dietary counselling — The dietary counseling will be delivered to mothers through group sessions (will include cooking demonstration) and home visits by lay health workers. The counseling will promote foods that are nutritious and locally available and general better food preparation practices. The choices of the foods to be promoted will be based on linear programming results from a preceding survey on dietary intake of pregnant women in the area as well as results of analysis of foods associated with infant birth size (same data). The goal in the linear programming was to find a model of food combinations among the most frequently consumed foods which better meets required intakes during pregnancy. Additionally, adherence to pregnancy iron supplements will also be promoted.
  Arms: Intervention
Behavioral: Community based antenatal counselling — The antenatal counselling will focus on preparations for neonatal care and encouragement for facility based delivery.

SUMMARY:
High neonatal mortality rates accounts for a substantial early loss of lives in Malawi; and has thus been a hindrance for Malawi to eradicate child deaths. From 2000 to 2011, Malawi achieved an overall reduction of 23% in under-five child mortality. The reduction was more substantial between the second and the fifth year of life, being 28%. However, in the neonatal period the reduction was half, at 14%. Neonatal deaths in developing countries are due to prematurity or low birth weight, neonatal infections, birth trauma related conditions and congenital anomalies.

Being of low birth weight increases the risk of death four fold in the neonatal period. Even when low birth weight infants survive, their poorly developed immune function exposes them to increased morbidity in early life. Maternal nutrition represents by far the greatest influence among pregnancy environmental on birth weight in low income countries. There is strong evidence that health and dietary counselling is effective in improving child nutrition outcomes. Thus we propose to test the effectiveness in improving birth weight by a low cost intervention, community based health and nutrition counselling delivered to mothers during pregnancy in Malawi.

On the other hand, in the Malawian context offering individualized dietetic counselling could be impeded by the healthcare workforce short fall. Currently the health workforce does not include dieticians . The use of lay health workers (LHW) has been identified as one of the effective strategies to meet the health workforce shortage challenges in low resource settings.

It is on this basis that a study was planned, aimed at developing lay health worker delivered community based nutrition counselling to mothers during pregnancy and measuring its effectiveness in improving birth weight in the Malawian context. The study was comprised of an initial i) formative study, followed by ii) a cross-sectional survey. Findings of these two sub-studies were utilized to develop a nutrition counselling intervention. Finally iii) a cluster Randomized Controlled Trial (cRCT) aimed at measuring the effect of the intervention on birth size (weight, length, arm and abdominal circumferences) will now be conducted which is being elaborated in this protocol.

DETAILED DESCRIPTION:
High neonatal mortality rates accounts for a substantial early loss of lives in Malawi; and has thus been a hindrance for Malawi to eradicate child deaths. From 2000 to 2011, Malawi achieved an overall reduction of 23% in under-five child mortality. The reduction was more substantial between the second and the fifth year of life, being 28%. However, in the neonatal period the reduction was half, at 14%. Neonatal deaths in developing countries are due to prematurity or low birth weight, neonatal infections, birth trauma related conditions and congenital anomalies.

Being of low birth weight increases the risk of death four fold in the neonatal period. Even when low birth weight infants survive, their poorly developed immune function exposes them to increased morbidity in early life. Maternal nutrition represents by far the greatest influence among pregnancy environmental on birth weight in low income countries. There is strong evidence that health and dietary counselling is effective in improving child nutrition outcomes. Thus we propose to test the effectiveness in improving birth weight by a low cost intervention, community based health and nutrition counselling delivered to mothers during pregnancy in Malawi.

On the other hand, in the Malawian context offering individualized dietetic counselling could be impeded by the healthcare workforce short fall. Currently the health workforce does not include dieticians . The use of lay health workers (LHW) has been identified as one of the effective strategies to meet the health workforce shortage challenges in low resource settings.

It is on this basis that a study was planned, aimed at developing lay health worker delivered community based nutrition counselling to mothers during pregnancy and measuring its effectiveness in improving birth weight in the Malawian context. The study was comprised of an initial i) formative study, followed by ii) a cross-sectional survey. Findings of these two sub-studies were utilized to develop a nutrition counselling intervention. Finally iii) a cluster Randomized Controlled Trial (cRCT) aimed at measuring the effect of the intervention on birth size (weight, length, arm and abdominal circumferences) will now be conducted which is being elaborated in this protocol.

Three hundred pregnant women, at ≥12 weeks but ≤ 16 weeks of gestation, will be recruited from Nankumba Traditional Authority (TA) area, in Mangochi district. They will be offered community based dietary counselling aiming at improving dietary intake to meet their nutritional needs.

Measurement of study outcomes will be as follows: Infant birthweight will be collected at the end of the study while as dietary intake (including dietary perceptions), anthropometric status, and biochemical nutrition status will be assessed at enrollment, and two additional time points before the end point.

ELIGIBILITY:
Inclusion Criteria:

1. Pregnant at ≥ 6 weeks but ≤ 17 weeks of gestation
2. Available during the period of the study.
3. Intention to reside in the study area in the next 6 months
4. Intention to give birth at the health facilities within the study area
5. Consent to participate (indicated by a signature or fingerprint)

Exclusion Criteria:

1. Severe illness, where the mother is bed ridden
2. Multiple births

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 300 (Actual)
Dates: Start 2015-11-01 (Actual); Primary Completion 2017-04-12 (Actual); Study Completion 2017-12-31 (Actual)

PRIMARY OUTCOMES:
Infant birthweight | 1 hour
  Infant birthweight measured within an hour after birth

SECONDARY OUTCOMES:
Infant birth length | 1 hour
  Infant birth length measured within an hour after birth
Infant birth head circumference | 1 hour
  Infant head circumference measured within an hour after birth
Infant birth abdomen circumference | 1 hour
  Infant birth abdomen circumference measured within an hour after birth
Pregnancy body mass index | At 8-22 weeks; 35 weeks of gestation
  Weight, Height, during
Pregnancy blood glucose level | At 8-22 weeks; 35 weeks of gestation
  Blood glucose measured in milligram per decilitre
Pregnancy hemoglobin count | At 8-22 weeks; 35 weeks of gestation
  Hemoglobin count in grams per decilitre
Pregnancy skinfold thickness | At 8-22 weeks; 35 weeks of gestation
  Skinfold thicknesses (subscapular, biceps, triceps, suprailiac)
Pregnancy food intake | At 8-22 weeks; 35 weeks of gestation
  Quantified food intake past 24 hours
Knowledge of healthy foods | At 8-22 weeks; 35 weeks of gestation
  Perceptions towards food, eating habits

CONTACTS AND LOCATIONS:
Overall Officials: Penjani R Kamudoni, PhD, Principal Investigator — University of Oslo
Locations (1):
- Monkey bay community hospital, Mangochi, Malawi

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Kamudoni PR, Kaunda L, Tharrey M, Mphande M, Chithambo S, Ferguson E, Shi Z, Mdala I, Maleta K, Munthali A, Holmboe-Ottesen G, Iversen PO. Context-Tailored Food-Based Nutrition Education and Counseling for Pregnant Women to Improve Birth Outcomes: A Cluster-Randomized Controlled Trial in Rural Malawi. Curr Dev Nutr. 2024 Nov 7;8(12):104506. doi: 10.1016/j.cdnut.2024.104506. eCollection 2024 Dec. PMID 39654971
- [Derived] Katenga-Kaunda LZ, Iversen PO, Kamudoni PR, Holmboe-Ottesen G, Fjeld HE. Food-based nutrition counselling and education intervention for improved diets of pregnant women in rural Malawi: a qualitative study of factors influencing dietary behaviour change. Public Health Nutr. 2022 Sep;25(9):2436-2447. doi: 10.1017/S1368980022000593. Epub 2022 Apr 4. PMID 35369896
- [Derived] Katenga-Kaunda LZ, Kamudoni PR, Holmboe-Ottesen G, Fjeld HE, Mdala I, Shi Z, Iversen PO. Enhancing nutrition knowledge and dietary diversity among rural pregnant women in Malawi: a randomized controlled trial. BMC Pregnancy Childbirth. 2021 Sep 22;21(1):644. doi: 10.1186/s12884-021-04117-5. PMID 34551744
- [Derived] Ziyenda Katenga-Kaunda L, Iversen PO, Holmboe-Ottesen G, Fjeld H, Mdala I, Kamudoni PR. Dietary intake and processes of behaviour change in a nutrition education intervention for pregnant women in rural Malawi: a cluster-randomised controlled trial. Public Health Nutr. 2020 Sep;23(13):2345-2354. doi: 10.1017/S1368980020000294. Epub 2020 May 18. PMID 32419688